CLINICAL TRIAL: NCT04110665
Title: Evaluation of Multimodal Oral Strategies Using Sequential Analysis (Tramadol, Opioid) After Shoulder Ambulatory Surgery
Brief Title: Multimodal Analgesia Strategies After Major Shoulder Ambulatory Surgery
Acronym: Shoulder1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Local/2017/PC-03; 2017-A01316-47 (Other: ANSM)
Record Dates: First submitted 2019-09-10; First posted 2019-10-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Tendon Injuries
Keywords: shoulder; surgery; analgesia; opioid
MeSH Terms: conditions — Tendon Injuries; Agnosia | interventions — Tramadol; Acetaminophen; Nefopam; Morphine; Oxycodone

STUDY DESIGN:
Intervention Model Description: Evaluation of the treatment based on QoR40 survey every 20 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Paracetamol+ ketoprofene and Tramadol (Active Comparator): Paracetamol per os 1g every 6 hours and ketoprofene 100 mg per os every 12 hours were systematically administered. Tramadol 100 mg per os every 6 hours was added when pain was > 3/10 on a numeric ranking scale (0 no pain, 10 worst pain).
  Interventions: Drug: Tramadol
- Paracetamol+ ketoprofene+ Nefopam and Tramadol (Active Comparator): Paracetamol per os 1g every 6 hours and ketoprofene 100 mg per os every 12 hours and Nefopam 120 mg intravenously were systematically administered. Tramadol 100 mg per os every 6 hours was added when pain was > 3/10 on a numeric ranking scale (0 no pain, 10 worst pain).
  Interventions: Drug: Tramadol; Drug: Nefopam 20 MG/ML
- Paracetamol+ ketoprofene and morphine (Active Comparator): Paracetamol per os 1g every 6 hours and ketoprofene 100 mg per os every 12 hours were systematically administered. Opioid immediate release (morphine 10 mg) per os every 6 hours was added when pain was > 3/10 on a numeric ranking scale (0 no pain, 10 worst pain).
  Interventions: Drug: Morphine Sulfate
- Paracetamol+ ketoprofene+Opioid delayed release and morphine (Active Comparator): Paracetamol per os 1g every 6 hours and ketoprofene 100 mg per os every 12 hours and 20 mg of opioid delayed release (Oxycodone) were systematically administered. Opioid immediate release (morphine 10 mg) per os every 6 hours was added when pain was > 3/10 on a numeric ranking scale (0 no pain, 10 worst pain).
  Interventions: Drug: Morphine Sulfate; Drug: Oxycodone 20mg

INTERVENTIONS:
Drug: Tramadol — Tramadol 100 mg tablet
  Other Names: Paracetamol; Ketoprofene
  Arms: Paracetamol+ ketoprofene and Tramadol; Paracetamol+ ketoprofene+ Nefopam and Tramadol
Drug: Nefopam 20 MG/ML — 120 mg for 24 hours
  Other Names: Paracetamol; Ketoprofene; Tramadol
  Arms: Paracetamol+ ketoprofene+ Nefopam and Tramadol
Drug: Morphine Sulfate — Tablet 10mg
  Other Names: Paracetamol; Ketoprofene
  Arms: Paracetamol+ ketoprofene and morphine; Paracetamol+ ketoprofene+Opioid delayed release and morphine
Drug: Oxycodone 20mg — release
  Other Names: Paracetamol; Ketoprofene; Morphine Sulfate
  Arms: Paracetamol+ ketoprofene+Opioid delayed release and morphine

SUMMARY:
This study evaluates the addition of tramadol, or nefopam or opioid to paracetamol and ketoprofene in the treatment of pain in adults after shoulder ambulatory surgery. In a first step, 30 patients will receive tramadol as rescue analgesia in combination with paracetamol and ketoprofene, while the other will receive nefopam or opioid in a sequential analysis that will be performed every 20 patients using the QoR 40 survey.

DETAILED DESCRIPTION:
Multimodal analgesia using acetaminophen with non steroidal anti inflammatory is commonly used for pain relief after ambulatory surgery. Tramadol achieves pain relief when rescue analgesia is needed after this surgery, but induces side effects (nausea, vomiting, discomfort, sleep disorder...). Other drugs could be used to reduce the side effects of tramadol and improve postoperative experience : nefopam or opioid (immediate or delayed release medication). Using a survey that describes pain, comfort, emotion or physical status (QoR 40), the investigators analyse the impact of various multimodal strategies using tramadol or nefopam or opioid that is necessary to improve postoperative experience.

ELIGIBILITY:
Inclusion Criteria:

* shoulder surgery
* under general anesthesia with an nterscalenic block
* written informed consent
* age > 18 years

Exclusion Criteria:

* age < 18years
* emergency surgery
* refusal
* drug or opioid abuses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR) 40 survey | Day 2
  score based on 200 points (minimum 40, maximum 200), 40 questions (5 points for each question)

CONTACTS AND LOCATIONS:
Overall Officials: benjamin Garnaud, MD, Study Director — CHU Nimes, Nimes University, France
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garnaud B, Mares O, L'hermite J, Vialles N, Gricourt Y, Lannelongue A, Lefrant JY, Cuvillon P. Multimodal oral analgesia strategy after ambulatory arthroscopic shoulder surgery: case series using adaptive therapeutic approaches by sequential analysis. J Shoulder Elbow Surg. 2021 Feb;30(2):250-257. doi: 10.1016/j.jse.2020.08.040. Epub 2020 Sep 18. PMID 32950669